CLINICAL TRIAL: NCT03183934
Title: A Follow-up Study to Evaluate the Efficacy and Safety for the Patients With ALLO-ASC-DFU Treatment in Phase 1/2 Clinical Trial of ALLO-ASC-EB-101
Brief Title: A Follow-up Study to Evaluate the Efficacy and Safety of ALLO-ASC-DFU in ALLO-ASC-EB-101 Clinical Trial
Status: Completed | Type: Observational
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLO-ASC-EB-102
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Dystrophic Epidermolysis Bullosa
Keywords: Epidermolysis Bullosa; Stem cell
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: ALLO-ASC-DFU — ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor(VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a Dystrophic Epidermolysis Bullosa.
  This study is a follow-up study without intervention.
  Other Names:
  Allogenic adipose-derived mesenchymal stem cells

SUMMARY:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 1/2 clinical trial(ALLO-ASC-EB-101) for 24 months.

DETAILED DESCRIPTION:
This is an open-label follow up study to evaluate the efficacy and safety for the subjects with ALLO-ASC-DFU treatment in phase 1/2 clinical trial (ALLO-ASC-EB-101) for 24 months.

ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor(VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a Dystrophic Epidermolysis Bullosa.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are treated with ALLO-ASC-DFU sheet in phase 1/2 clinical trial of ALLO-ASC-EB-101.
2. A subject who is willing to follow the protocol and provide informed consent on screening, given that the information with respect to the clinical trial is provided.

Exclusion Criteria:

1. Subjects who are considered not suitable for the study by the principal investigator.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subject is enrolled who are treated with ALLO-ASC-DFU sheet in phase 1/2 clinical trial of ALLO-ASC-EB-101
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Safety assessed by clinically measured abnormality of laboratory tests and adverse events | Every time of visit for follow up to 24 months
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability.

SECONDARY OUTCOMES:
Area of re-epithelization | Every time of visit for follow up to 24 months
  Time taken to re-epithelization

CONTACTS AND LOCATIONS:
Overall Officials: Su Chan Kim, PhD, Principal Investigator — Gangnam Severence Hospital
Locations (1):
- Gangnam Severence Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No